CLINICAL TRIAL: NCT06841354
Title: A Phase 3, Randomized, Open-label Study Comparing Efficacy and Safety of Sacituzumab Tirumotecan (Sac-TMT, MK-2870) as a Monotherapy and in Combination With Pembrolizumab (MK-3475) Versus Treatment of Physician's Choice in Participants With Previously Untreated Locally Recurrent Unresectable or Metastatic Triple-Negative Breast Cancer Expressing PD-L1 at CPS Less Than 10 (TroFuse-011)
Brief Title: A Study of Sacituzumab Tirumotecan (Sac-TMT, MK-2870) as Monotherapy and in Combination With Pembrolizumab (MK-3475) in Participants With Triple-Negative Breast Cancer (MK-2870-011/TroFuse-011)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2870-011; MK-2870-011 (Other: MSD); TroFuse-011 (Other: MSD); 2024-516834-36-00 (Registry Identifier: EU CT); U1111-1311-2310 (Registry Identifier: UTN)
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Triple Negative Breast Neoplasms
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2); Antibody-drug conjugate (ADC); Trophoblast cell-surface antigen 2 (TROP2)
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Paclitaxel; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Sacituzumab Tirumotecan (Experimental): Participants receive sacituzumab tirumotecan intravenously (IV) at a dose of 4 mg/kg every 2 weeks (Q2W) until disease progression, toxicity or discontinuation.
  Interventions: Biological: Sacituzumab tirumotecan; Drug: Rescue Medication
- Arm B: Sacituzumab Tirumotecan + Pembrolizumab (Experimental): Participants receive sacituzumab tirumotecan IV 4 mg/kg Q2W until disease progression, toxicity or discontinuation PLUS pembrolizumab IV 400 mg every 6 weeks (Q6W) for up to 18 administrations (up to ~2 years).
  Interventions: Biological: Sacituzumab tirumotecan; Biological: Pembrolizumab; Drug: Rescue Medication
- Arm C: Treatment of Physician's Choice (TPC) (Active Comparator): Participants receive physician's choice of chemotherapy agent(s): paclitaxel IV 80 mg/m^2 once every week (Q1W) OR paclitaxel IV 90 mg/m^2 on Days 1, 8, and 15, every 4 weeks (Q4W) OR nab-paclitaxel IV 100 mg/m^2 on Days 1, 8, and 15, Q4W OR gemcitabine IV 1000 mg/m^2 on Days 1 and 8, every 3 weeks (Q3W) PLUS carboplatin IV area under the curve (AUC) 2 mg/mL/min on Days 1 and 8, Q3W, until disease progression, toxicity or discontinuation.
  Interventions: Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Biological: Sacituzumab tirumotecan — IV Infusion
  Other Names: Sac-TMT; MK-2870
  Arms: Arm A: Sacituzumab Tirumotecan; Arm B: Sacituzumab Tirumotecan + Pembrolizumab
Biological: Pembrolizumab — IV Infusion
  Other Names: MK-3475; Keytruda®
  Arms: Arm B: Sacituzumab Tirumotecan + Pembrolizumab
Drug: Rescue Medication — Participants receive the following pre-medications before sacituzumab tirumotecan infusion: Histamine-1 (H1) receptor agonist, histamine-2 (H2) receptor antagonist, acetaminophen or equivalent, dexamethasone or equivalent infusion. Participants are also recommended to receive prophylactic steroid mouthwash (dexamethasone or equivalent).
  Arms: Arm A: Sacituzumab Tirumotecan; Arm B: Sacituzumab Tirumotecan + Pembrolizumab
Drug: Paclitaxel — IV Infusion
  Other Names: Taxol; Onxol
  Arms: Arm C: Treatment of Physician's Choice (TPC)
Drug: Nab-paclitaxel — IV Infusion
  Other Names: Abraxane
  Arms: Arm C: Treatment of Physician's Choice (TPC)
Drug: Gemcitabine — IV Infusion
  Other Names: Gemzar
  Arms: Arm C: Treatment of Physician's Choice (TPC)
Drug: Carboplatin — IV Infusion
  Other Names: Paraplatin
  Arms: Arm C: Treatment of Physician's Choice (TPC)

SUMMARY:
Researchers want to know if sacituzumab tirumotecan given alone or with pembrolizumab can treat triple negative breast cancer (TNBC). The main goal of this study is to learn if people treated with sacituzumab tirumotecan alone or with pembrolizumab live longer overall or without the cancer growing or spreading compared to people treated with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has locally recurrent unresectable or metastatic TNBC that cannot be treated with curative intent
* Has not received systemic treatment for locally recurrent unresectable or metastatic breast cancer
* Participants previously treated for early-stage breast cancer must have completed all prior therapy for early-stage breast cancer with curative intent at least 6 months before the first disease recurrence
* Is a candidate for treatment with pembrolizumab and one of the TPC options: paclitaxel or nab-paclitaxel or gemcitabine + carboplatin
* Participants who have AEs due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline with the exception of alopecia or vitiligo. Participants with endocrine-related AEs who are adequately treated with hormone replacement are eligible
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks, and have undetectable HBV viral load
* Participants with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has breast cancer amenable to treatment with curative intent
* Has TNBC with evaluable tumor programmed death ligand 1 (PD-L1) expression at combined positive score (CPS) ≥10
* Has received prior systemic therapy for treatment of locally recurrent unresectable or metastatic breast cancer
* Has Grade ≥2 peripheral neuropathy
* Has history of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or severe corneal disease that prevents/delays corneal healing
* Has active inflammatory bowel disease requiring immunosuppressive medication or previous history of inflammatory bowel disease
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease
* Has skin only metastatic disease
* Has advanced/metastatic, symptomatic visceral spread at risk of rapidly evolving into life-threatening complications
* Human immunodeficiency virus (HIV)-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has known additional malignancy that is progressing or has required active treatment within the past 5 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable
* Active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid) is allowed
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV deoxyribonucleic acid (DNA)) and Hepatitis C virus (HCV) (defined as anti-HCV antibody (Ab) positive and detectable HCV ribonucleic acid (RNA)) infection
* History of stem cell/solid organ transplant
* Has not adequately recovered from major surgery or has ongoing surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-16 (Actual); Primary Completion 2030-05-18 (Estimated); Study Completion 2030-05-18 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) (sac-TMT versus treatment of physician's choice (TPC); sac-TMT plus pembrolizumab versus TPC) | Up to ~37 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) based on blinded independent central review (BICR) or death due to any cause, whichever occurs first. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD.
Overall Survival (OS) (sac-TMT versus TPC) | Up to ~61 months
  OS is defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) (sac-TMT plus pembrolizumab versus treatment of physician's choice (TPC); sac-TMT plus pembrolizumab versus sac-TMT) | Up to ~61 months
  OS is defined as the time from randomization to death due to any cause.
Progression-Free Survival (PFS) (sac-TMT plus pembrolizumab versus sac-TMT) | Up to ~37 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 based on BICR or death due to any cause, whichever occurs first. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD.
Objective Response Rate (ORR) (sac-TMT versus TPC; sac-TMT plus pembrolizumab versus TPC) | Up to ~37 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 based on BICR.
Duration of Response (DOR) | Up to ~37 months
  For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 based on BICR, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death, whichever occurs first. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD.
Change from baseline in global health status/quality of life scores, on the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) (sac-TMT versus TPC; sac-TMT plus pembrolizumab versus TPC) | Baseline and up to ~61 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status.
Change from baseline in physical functioning score, on the EORTC QLQ-C30 (sac-TMT versus TPC; sac-TMT plus pembrolizumab versus TPC) | Baseline and up to ~61 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better level of physical functioning.
Change from baseline in emotional functioning score, on the EORTC QLQ-C30 (sac-TMT versus TPC; sac-TMT plus pembrolizumab versus TPC) | Baseline and up to ~61 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to questions about their emotional functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better level of emotional functioning.
Change from baseline in fatigue score, on the EORTC QLQ-C30 (sac-TMT versus TPC; sac-TMT plus pembrolizumab versus TPC) | Baseline and up to ~61 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to questions about their fatigue are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better level of function.
Change from baseline in diarrhea score, on the EORTC QLQ-C30 (sac-TMT versus TPC; sac-TMT plus pembrolizumab versus TPC) | Baseline and up to ~61 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the question "Have you had diarrhea?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better level of function.
Number of participants who experience one or more adverse events (AEs) | Up to ~61 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants who discontinue study treatment due to an AE | Up to ~61 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (238):
- United States (35):
  - USA Mitchell Cancer Institute ( Site 0090), Mobile, Alabama
  - Ironwood Cancer & Research Centers ( Site 0036), Chandler, Arizona
  - City of Hope ( Site 0097), Duarte, California
  - City of Hope Lennar Foundation Cancer Center ( Site 0099), Irvine, California
  - UCLA Department of Medicine - Hematology & Oncology ( Site 0047), Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center ( Site 0016), San Francisco, California
  - Yale New Haven Hospital ( Site 0001), New Haven, Connecticut
  - Washington Hospital Center ( Site 0098), Washington D.C., District of Columbia
  - AdventHealth Medical Group Oncology and Hematology at Altamonte ( Site 0007), Altamonte Springs, Florida
  - Florida Cancer Specialists - East ( Site 7000), West Palm Beach, Florida
  - University Cancer & Blood Center, LLC ( Site 0023), Athens, Georgia
  - St. Luke's Cancer Institute: Boise ( Site 0037), Boise, Idaho
  - University of Illinois Cancer Center ( Site 0044), Chicago, Illinois
  - MedStar Franklin Square Medical Center ( Site 0031), Baltimore, Maryland
  - MedStar Good Samaritan Hospital ( Site 0079), Baltimore, Maryland
  - MedStar Montgomery Medical Center ( Site 0078), Olney, Maryland
  - Holy Cross Hospital ( Site 0091), Silver Spring, Maryland
  - Allina Health Cancer Institute ( Site 0069), Minneapolis, Minnesota
  - Comprehensive Cancer Centers of Nevada ( Site 0015), Las Vegas, Nevada
  - Renown Regional Medical Center ( Site 0005), Reno, Nevada
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0082), Hackensack, New Jersey
  - New Mexico Oncology Hematology Consultants Ltd. ( Site 0019), Albuquerque, New Mexico
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island ( Site 0073), Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center ( Site 0003), New York, New York
  - UNC REX Cancer Center ( Site 0071), Raleigh, North Carolina
  - SCRI Oncology Partners ( Site 7004), Nashville, Tennessee
  - Tennessee Oncology ( Site 0018), Nashville, Tennessee
  - Texas Oncology - DFW ( Site 8007), Dallas, Texas
  - Texas Oncology - West Texas ( Site 8004), El Paso, Texas
  - Kelsey Research Foundation ( Site 0040), Houston, Texas
  - Kelsey-Seybold Clinic - North Houston Campus ( Site 0096), Houston, Texas
  - Texas Oncology - San Antonio ( Site 8001), San Antonio, Texas
  - University of Utah, Huntsman Cancer Institute ( Site 0056), Salt Lake City, Utah
  - Virginia Oncology Associates (VOA) ( Site 8002), Norfolk, Virginia
  - Fred Hutchinson Cancer Center ( Site 0042), Seattle, Washington
- Argentina (7):
  - Instituto de Investigaciones Clinicas Mar del Plata ( Site 2401), Mar del Plata, Buenos Aires
  - Instituto Alexander Fleming ( Site 2402), Mar del Plata, Buenos Aires
  - Hospital Italiano de Cordoba ( Site 2406), Córdoba, Córdoba Province
  - Clinica Viedma ( Site 2403), Viedma, Río Negro Province
  - Fundacion Estudios Clinicos ( Site 2405), Rosario, Santa Fe Province
  - Hospital Provincial del Centenario ( Site 2410), Rosario, Santa Fe Province
  - Fundacion Centro Oncologico de Integración Regional ( Site 2400), Mendoza
- Australia (2):
  - Blacktown Hospital ( Site 5500), Blacktown, New South Wales
  - Peninsula Health Frankston Hospital ( Site 5501), Frankston, Victoria
- Belgium (4):
  - ZAS Sint Augustinus ( Site 3102), Antwerp, Flanders
  - Ziekenhuis Oost Limburg ( Site 3105), Genk, Limburg
  - AZ Maria Middelares ( Site 3103), Ghent, Oost-Vlaanderen
  - UZ Gent ( Site 3101), Ghent, Oost-Vlaanderen
- Brazil (6):
  - Hospital de Câncer de Recife ( Site 2300), Recife, Pernambuco
  - Liga Norte Riograndense Contra o Cancer ( Site 2310), Natal, Rio Grande do Norte
  - Hospital Nossa Senhora da Conceição ( Site 2302), Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII - Hospital de Cancer de Barretos ( Site 2307), Barretos, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto ( Site 2301), São Jose Do Rio Preto, São Paulo
  - IBCC - Núcleo de Pesquisa e Ensino ( Site 2306), São Paulo
- Canada (11):
  - Cross Cancer Institute ( Site 0216), Edmonton, Alberta
  - Lakeridge Health ( Site 0217), Oshawa, Ontario
  - North York General Hospital ( Site 0209), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0202), Toronto, Ontario
  - CIUSSS- saguenay-Lac-Saint-Jean ( Site 0213), Chicoutimi, Quebec
  - Centre Hospitalier de l'Université de Montréal ( Site 0208), Montreal, Quebec
  - Jewish General Hospital ( Site 0203), Montreal, Quebec
  - St. Marys Hospital Center ( Site 0201), Montreal, Quebec
  - McGill University Health Centre ( Site 0204), Montreal, Quebec
  - Hopital Du Saint-Sacrement ( Site 0210), Québec, Quebec
  - Saskatoon Cancer Centre ( Site 0215), Saskatoon, Saskatchewan
- Chile (6):
  - IC La Serena Research ( Site 2007), La Serena, Coquimbo Region
  - FALP ( Site 2000), Santiago, Region M. de Santiago
  - Clínica UC San Carlos de Apoquindo ( Site 2008), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 2001), Santiago, Region M. de Santiago
  - ONCOCENTRO APYS ( Site 2005), Viña del Mar, Región de Valparaíso
  - Biocenter ( Site 2009), Concepción, Región del Biobío
- China (23):
  - The First Afflilated Hospital of Bengbu Medical College ( Site 5022), Bengbu, Anhui
  - The First Affiliated Hospital of Chongqing Medical University ( Site 5039), Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Hospital ( Site 5020), Chongqing, Chongqing Municipality
  - The First Affiliated hospital of Xiamen University ( Site 5035), Xiamen, Fujian
  - Sun Yat-Sen University Cancer Center ( Site 5014), Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital. ( Site 5008), Nanning, Guangxi
  - Henan Cancer Hospital ( Site 5001), Zhengzhou, Henan
  - Tongji Hospital Tongji Medical Science & Technology ( Site 5007), Wuhan, Hubei
  - Xiangyang Central Hospital ( Site 5017), Xiangyang, Hubei
  - Jiangsu Province Hospital ( Site 5009), Nanjing, Jiangsu
  - Xuzhou Central Hospital ( Site 5036), Xuzhou, Jiangsu
  - The First Hospital of Jilin University ( Site 5003), Changchun, Jilin
  - The First Affiliated Hospital of Xi an Jiaotong University ( Site 5005), Xi'an, Shaanxi
  - Jinan Central Hospital ( Site 5031), Jinan, Shandong
  - LinYi Cancer Hospital ( Site 5021), Linyi, Shandong
  - Shanxi Cancer Hospital ( Site 5043), Taiyuan, Shanxi
  - Sichuan Cancer Hospital. ( Site 5018), Chengdu, Sichuan
  - The Second People's Hospital of Neijiang ( Site 5016), Neijiang, Sichuan
  - Affiliated Tumor Hospital of Xinjiang Medical University ( Site 5006), Ürümqi, Xinjiang
  - The First Affiliated Hospital Zhejiang University School of Medicine ( Site 5026), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 5012), Hangzhou, Zhejiang
  - The Second Affiliated hospital of Zhejiang University school of medicine ( Site 5024), Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province ( Site 5029), Linhai, Zhejiang
- Colombia (5):
  - Instituto de Cancerología ( Site 2206), Medellín, Antioquia
  - Centro Cancerologico del Caribe LTD ( Site 2209), Barranquilla, Atlántico
  - FUNDACION CTIC CENTRO DE TRATAMIENTO E INVESTIGACION SOBRE CANCER LUIS CARLOS SARMIENTO ANGULO ( Site 2203), Bogotá, Bogota D.C.
  - IMAT S.A.S ( Site 2202), Montería, Departamento de Córdoba
  - Oncologos Del Occidente ( Site 2208), Pereira, Risaralda Department
- Czechia (4):
  - Vseobecna fakultni nemocnice v Praze ( Site 3501), Prague, Praha 2
  - Masarykuv onkologicky ustav ( Site 3500), Brno, South Moravian
  - Fakultni nemocnice Olomouc ( Site 3502), Olomouc
  - Fakultni Thomayerova nemocnice ( Site 3506), Prague
- Denmark (4):
  - Rigshospitalet University Hospital ( Site 3201), Copenhagen, Capital Region
  - Herlev og Gentofte Hospital. ( Site 3205), Copenhagen, Capital Region
  - Aarhus Universitets hospital ( Site 3204), Aarhus, Central Jutland
  - Odense Universitetshospital ( Site 3202), Odense, Region Syddanmark
- Finland (3):
  - Oulun yliopistollinen sairaala-Oncology and Hematology ( Site 3304), Oulu, North Ostrobothnia
  - Tampereen yliopistollinen sairaala-Oncology ( Site 3302), Tampere, Pirkanmaa
  - Helsinki University Hospital - Comprehensive Cancer Center (HYKS - Syöpäkeskus) ( Site 3301), Helsinki, Uusimaa
- France (9):
  - CENTRE LEON BERARD ( Site 3004), Lyon, Auvergne-Rhône-Alpes
  - Clinique Francois Chenieux ( Site 3006), Limoges, Haute-Vienne
  - Institut Regional du Cancer Montpellier ( Site 3009), Montpellier, Herault
  - Institut De Cancerologie De L Ouest ( Site 3003), Saint-Herblain, Loire-Atlantique
  - Institut Jean Godinot ( Site 3002), Reims, Marne
  - Centre Henri Becquerel ( Site 3001), Rouen, Seine-Maritime
  - HIA Sainte Anne ( Site 3007), Toulon, Var
  - Groupe Hospitalier Paris Saint Joseph ( Site 3010), Paris
  - Hôpital Européen Georges Pompidou ( Site 3011), Paris
- Germany (5):
  - Universitatsklinikum Erlangen ( Site 4302), Erlangen, Bavaria
  - Luisenkrankenhaus Düsseldorf ( Site 4305), Düsseldorf, North Rhine-Westphalia
  - Kliniken Essen-Mitte, Evangelische Huyssens-Stiftung-Klinik für Senologie/ Brustzentrum ( Site 4304), Essen, North Rhine-Westphalia
  - Caritas Klinikum Saarbruecken St. Theresia ( Site 4301), Saarbrücken, Saarland
  - HELIOS Klinikum Berlin-Buch ( Site 4303), Berlin
- Greece (4):
  - Aretaieio Hospital ( Site 3900), Athens, Attica
  - University General Hospital of Heraklion-Internal Medicine-Oncology ( Site 3903), Heraklion, Irakleio
  - General University Hospital of Larissa, Oncology Clinic ( Site 3902), Larissa, Thessaly
  - European Interbalkan Medical Center ( Site 3901), Thessaloniki
- Hungary (3):
  - Békés Vármegyei Központi Kórház Pándy Kálmán Tagkórház-Megyei Onkológiai Centrum ( Site 3405), Gyula, Bekes County
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ-Onkoterapias Klinika ( Site 3407), Szeged, Csongrád megye
  - Budapesti Uzsoki Utcai Kórház-Onkoradiológiai Osztály ( Site 3408), Budapest, Pest County
- Israel (5):
  - Rambam Health Care Campus ( Site 3700), Haifa
  - Shaare Zedek Medical Center ( Site 3704), Jerusalem
  - Rabin Medical Center ( Site 3702), Petah Tikva
  - Sheba Medical Center ( Site 3701), Ramat Gan
  - Sourasky Medical Center ( Site 3703), Tel Aviv
- Italy (7):
  - Istituto Nazionale Tumori Regina Elena ( Site 4607), Rome, Roma
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola ( Site 4605), Bologna
  - Ospedale Policlinico San Martino ( Site 4606), Genova
  - IRCCS Ospedale San Raffaele ( Site 4600), Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 4601), Milan
  - Azienda Ospedaliero Universitaria Maggiore della Carità ( Site 4604), Novara
  - Policlincio Gemelli ( Site 4602), Roma
- Japan (21):
  - Aichi Cancer Center ( Site 5117), Nagoya, Aichi-ken
  - Nagoya City University Hospital ( Site 5108), Nagoya, Aichi-ken
  - National Hospital Organization Shikoku Cancer Center ( Site 5122), Matsuyama, Ehime
  - Hokkaido University Hospital ( Site 5100), Sapporo, Hokkaido
  - Tokai University Hospital ( Site 5107), Isehara, Kanagawa
  - Kanagawa Cancer Center ( Site 5106), Yokohama, Kanagawa
  - Mie University Hospital ( Site 5109), Tsu, Mie-ken
  - The University of Osaka Hospital ( Site 5111), Suita, Osaka
  - Saitama Medical University International Medical Center ( Site 5116), Hidaka, Saitama
  - Juntendo University Hospital ( Site 5104), Bunkyo, Tokyo
  - Cancer Institute Hospital of JFCR ( Site 5102), Koto, Tokyo
  - Showa Medical University Hospital ( Site 5103), Shinagawa, Tokyo
  - Tokyo Medical University Hospital ( Site 5121), Shinjuku, Tokyo
  - National Center for Global Health and Medicine ( Site 5105), Shinjuku, Tokyo
  - Akita University Hospital ( Site 5115), Akita
  - Fukushima Medical University Hospital ( Site 5101), Fukushima
  - Hiroshima City Hiroshima Citizens Hospital ( Site 5113), Hiroshima
  - Social medical corporation Hakuaikai Sagara Hospital ( Site 5114), Kagoshima
  - Kyoto University Hospital ( Site 5110), Kyoto
  - Okayama University Hospital ( Site 5118), Okayama
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute ( Site 5112), Osaka
- Malaysia (4):
  - National Cancer Institute ( Site 5401), Putrajaya, Putrajaya
  - Sarawak General Hospital ( Site 5400), Kuching, Sarawak
  - Pantai Hospital Kuala Lumpur ( Site 5402), Kuala Lumpur
  - University Malaya Medical Centre ( Site 5403), Kuala Lumpur
- Mexico (11):
  - CIO - Centro de Inmuno-Oncología de Occidente ( Site 2504), Guadalajara, Jalisco
  - Grupo Médico ASSET ( Site 2507), Mexico City, Mexico City
  - COI Centro Oncologico Internacional S.A.P.I. de C.V. ( Site 2514), Mexico City, Mexico City
  - Centro Oncologico de Alta Especialidad, S.C. ( Site 2509), Mexico City, Mexico City
  - Higiea Oncologia ( Site 2505), Mexico City, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez" ( Site 2501), Monterrey, Nuevo León
  - Oncare - Unidad Valle ( Site 2502), San Pedro Garza García, Nuevo León
  - Centro de Investigacion Clinica de Oaxaca ( Site 2503), Oaxaca City, Oaxaca
  - Centro de Investigación Oncológica Galerías SC ( Site 2511), Aguascalientes
  - Unidad de Mastologia Avanzada de Chihuahua S.A de C.V ( Site 2510), Chihuahua City
  - Centro Potosino de Investigación Médica ( Site 2512), San Luis Potosí City
- Netherlands (6):
  - Ziekenhuis Rijnstate ( Site 4501), Arnhem, Gelderland
  - Zuyderland Medical Centre ( Site 4507), Sittard Geleen, Limburg
  - ETZ Elisabeth ( Site 4504), Tilburg, North Brabant
  - Deventer Ziekenhuis ( Site 4503), Deventer, Overijssel
  - Erasmus Medisch Centrum ( Site 4505), Rotterdam, South Holland
  - Meander Medisch Centrum ( Site 4500), Amersfoort, Utrecht
- New Zealand (2):
  - Harbour Cancer & Wellness ( Site 5600), Newmarket, Auckland
  - Bowen Hospital ( Site 5601), Wellington
- Peru (4):
  - Clínica Internacional - Sede San Borja ( Site 2604), Lima
  - IPOR Instituto Peruano de Oncología & Radioterapia ( Site 2601), Lima
  - Oncosalud ( Site 2600), Lima
  - Hospital Militar Central Coronel Luis Arias Schereiber ( Site 2603), Lima
- Philippines (2):
  - Mary Mediatrix Medical Center ( Site 5702), Lipa, Batangas
  - THE MEDICAL CITY ILOILO ( Site 5704), Iloilo City
- Poland (8):
  - Wielkopolskie Centrum Onkologii-Oddział Onkologii Klinicznej i Immunoonkologii z Pododdziałem Dzien ( Site 3811), Poznan, Greater Poland Voivodeship
  - Centrum Onkologii im prof Franciszka Lukaszczyka ( Site 3802), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Pratia MCM Krakow ( Site 3812), Krakow, Lesser Poland Voivodeship
  - Mazowiecki Szpital Wojewódzki w Siedlcach-Siedleckie Centrum Onkologii ( Site 3801), Siedlce, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworów Piersi i Chirurgii ( Site 3803), Warsaw, Masovian Voivodeship
  - Mazowiecki Szpital Onkologiczny ( Site 3807), Wieliszew, Masovian Voivodeship
  - Szpitale Pomorskie Sp. z o. o. ( Site 3805), Gdynia, Pomeranian Voivodeship
  - Szpital Wojewodzki im.M.Kopernika. ( Site 3800), Koszalin, West Pomeranian Voivodeship
- Romania (7):
  - Institutul Oncologic Cluj ( Site 4701), Cluj-Napoca, Cluj
  - S.C. Radiotherapy Center Cluj S.R.L ( Site 4705), Comuna Floresti, Cluj
  - Centrul de Oncologie "Sfântul Nectarie" ( Site 4702), Craiova, Dolj
  - Spitalul Municipal Schuller Ploiești ( Site 4707), Ploieşti, Prahova
  - Cabinet Medical Oncomed ( Site 4704), Timișoara, Timiș County
  - Spitalul Clinic Filantropia ( Site 4703), Bucharest
  - Centrul Medical Neolife- Baneasa ( Site 4706), Bucharest
- South Korea (6):
  - National Cancer Center ( Site 5202), Goyang-si, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 5204), Seongnam, Kyonggi-do
  - Kyungpook National University Chilgok Hospital ( Site 5205), Daegu, Kyongsangbuk-do
  - Seoul National University Hospital ( Site 5200), Seoul
  - Severance Hospital Yonsei University Health System ( Site 5201), Seoul
  - Samsung Medical Center ( Site 5203), Seoul
- Spain (7):
  - HOSPITAL UNIVERSITARIO VIRGEN DEL ROCIO-Medical Oncology ( Site 4104), Seville, Andalusia
  - ICO L Hospitalet ( Site 4101), L'Hospitalet de Llobregat, Barcelona
  - Hospital Clinico San Carlos ( Site 4100), Madrid, Madrid, Comunidad de
  - Hospital General Universitario de Valencia ( Site 4102), Valencia, Valenciana, Comunitat
  - Parc de Salut Mar - Hospital del Mar ( Site 4106), Barcelona
  - Hospital Beata María Ana ( Site 4105), Madrid
  - Hospital Universitario Ramon y Cajal ( Site 4103), Madrid
- Taiwan (5):
  - Taichung Veterans General Hospital ( Site 5303), Taichung
  - National Cheng Kung University Hospital ( Site 5304), Tainan
  - National Taiwan University Hospital ( Site 5300), Taipei
  - Mackay Memorial Hospital ( Site 5301), Taipei
  - Chang Gung Memorial Hospital ( Site 5302), Taoyuan District
- Thailand (3):
  - Faculty of Medicine Siriraj Hospital ( Site 5800), Bangkoknoi, Bangkok
  - Songklanagarind hospital ( Site 5801), Hat Yai, Changwat Songkhla
  - Faculty of Medicine - Khon Kaen University ( Site 5802), Khon Kaen
- Turkey (Türkiye) (4):
  - Adana Medical Park Seyhan Hastanesi ( Site 4804), Adana
  - Hacettepe Universite Hastaneleri ( Site 4800), Ankara
  - Sakarya Egitim Arastirma Hsatanesi ( Site 4809), Sakarya
  - Samsun Medical Park Hastanesi ( Site 4810), Samsun
- United Kingdom (5):
  - Royal Cornwall Hospital ( Site 4003), Truro, Cornwall
  - St Bartholomew's Hospital ( Site 4001), London, London, City of
  - University College London Hospital ( Site 4007), London, London, City of
  - Nottingham University Hospital NHS Trust ( Site 4009), Nottingham, Nottinghamshire
  - St. James s University Hospital ( Site 4004), Leeds

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/